CLINICAL TRIAL: NCT05328271
Title: A Pilot Study to Determine the Bioavailability of Oral Beta-Aminoisobutyric Acid (BAIBA) Ingestion
Acronym: BBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Collaborators: NNB Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB-21-34
Record Dates: First submitted 2022-03-29; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Absorption; Chemicals
MeSH Terms: interventions — 3-aminoisobutyric acid

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, crossover design
Who Masked: Participant, Investigator
Masking Description: Supplements blinded to participant and investigator by third party
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Beta-Aminoisobutyric Acid
- 1500 mg L-Valine (Active Comparator): 1500 mg L-Valine
  Interventions: Dietary Supplement: Beta-Aminoisobutyric Acid
- 250 mg Beta-Aminoisobutryic Acid (Experimental): 250 mg Beta-Aminoisobutryic Acid
  Interventions: Dietary Supplement: Beta-Aminoisobutyric Acid
- 500 mg Beta-Aminoisobutryic Acid (Experimental): 500 mg Beta-Aminoisobutryic Acid
  Interventions: Dietary Supplement: Beta-Aminoisobutyric Acid
- 1500 mg Beta-Aminoisobutryic Acid (Experimental): 1500 mg Beta-Aminoisobutryic Acid
  Interventions: Dietary Supplement: Beta-Aminoisobutyric Acid

INTERVENTIONS:
Dietary Supplement: Beta-Aminoisobutyric Acid — All supplements provided to all research participants containing BAIBA, L-Valine or placebo will be procured and prepared in a similar manner. Briefly, beta-amino isobutyric acid (BAIBA), L-Valine (an amino acid), and a resistant starch commonly consumed in various foods will be used as test agents for this study protcol. All supplements (both BAIBA and Valine) as well as placebo are produced and provided by NNB Nutrition. A certificate of analysis is provided in the attachments for the BAIBA. All supplements (BAIBA, L-Valine, and placebo) will be administered in gelatin capsules and consumed with a specified amount of cold tap water. The same number of capsules will be administered each time. All doses will be capsulated by manufacturer prior to use in the study protocol.

SUMMARY:
Think of this section as your research "elevator pitch." Please briefly describe the question(s) or issues you are addressing with your research (limited to 100 words). You will be able to provide information on specific outcomes, hypothesis, or related analysis in a following question.

Beta-amino isobutyric acid (BAIBA) is a myokine produced in skeletal muscle and has been shown to impact how our body metabolizes fuel. We seek to determine the bioavailability of different doses of orally ingested beta-aminoisobutyric acid (BAIBA).

DETAILED DESCRIPTION:
Once determined eligible and provided consent, participants will be assigned in a randomized, double-blind, placebo-controlled, crossover fashion. Eligible study participants will complete one of five testing conditions outlined below. For each testing condition, study participants will arrive in the lab after observing an overnight fast. Upon arrival, participants will donate the first of seven venous blood samples. Follow-up blood samples will be collected at 30, 60, 90, 120, 240, 300 minutes. The first and last collected samples will be collected into one 8mL SST and three 4mL EDTA tubes, while the second, third, and forth collected samples will be into two 4mL EDTA tubes, and have aliquots of 600 ul of plasma isolated and frozen at -80oC. Collected plasma will be analyzed for changes in beta-aminoisobutyric acid (BAIBA) and biomarkers commonly assessed by physicians to evaluate healthy. Participants will observe a minimum of 48 hours washout between conditions.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be between the ages of 18-50 years
* All participants will be required to abstain from taking any amino acid (i.e., BCAAs, creatine, - beta-alanine, carnitine, etc.) for 14 days prior to beginning this study and for the entire duration -of the study
* Body mass index between 18.5 - 29.9 kg/m2
* Report accumulating at least 30 minutes of physical activity three days per week
* All participants will be determined to be healthy through completion of a detailed health history questionnaires

Exclusion Criteria:

* Are less than 18 or greater than 50 years of age. Participants younger than 18 are excluded due to necessity of parental consent. Participants greater than 50 years old are excluded due to the anticipated age-related changes that occur in digestive function, medication use, and other - associated confounding comorbidities.
* Have a body mass index < 18.5 and > 29.9 kg/m2. Any participant with a BMI > 29.9 kg/m2 must have a body fat percentage below 30% to be eligible.
* No individuals with a BMI above 32.0 kg/m2 will be eligible, irrespective of their body composition.
* Have a fasting capillary glucose (-30 minutes) level > 110 mg/dL on two separate occasions.
* Currently smoke or have quit smoking within the past six months
* Are currently following a ketogenic diet or a very low-carbohydrate diet for the past 30 days.
* Any individual who is currently being treated for or diagnosed with a cardiac, respiratory, circulatory, musculoskeletal, metabolic, obesity, immune, autoimmune, psychiatric, hematological, neurological or endocrinological disorder or disease will be excluded.
* Report accumulating less than 30 minutes of physical activity per day for at least three days per week.
* Do not or are not willing to abstain from alcohol, nicotine and caffeine for 12 hours prior to each visit will be excluded
* Do not or are not willing to abstain from exercise for 24 hours prior to each visit will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of BAIBA. | 4 hours
  Plasma concentrations of BAIBA.

SECONDARY OUTCOMES:
Complete Blood Count | 4 hours
  Plasma and serum indicators of health
Comprehensive Metabolic Panel | 4 hours
  Plasma and serum indicators of health
Adverse Events | 4 hours
  Incidence and associations of reported adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Lindenwood University, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krieger JM, Hagele AM, Orr LS, Walden KE, Gross KN, Mumford PW, Kerksick CM. Dose-Response Absorption Kinetics of Oral L-Beta-Aminoisobutyric Acid (L-BAIBA) Supplementation in Healthy Men and Women. J Diet Suppl. 2023;20(6):832-849. doi: 10.1080/19390211.2022.2128141. Epub 2022 Oct 2. PMID 36184601